CLINICAL TRIAL: NCT00629135
Title: Single Centre, Prospective, Comparative, Open-label, Randomised Study to Evaluate the Efficacy and Tolerability of the Combination of Moxifloxacin Plus Metronidazole Versus Piperacillin/Tazobactam for the Treatment of Patients With Intra-abdominal Abscesses
Brief Title: Moxifloxacin Plus Metronidazole Versus Piperacillin/Tazobactam for the Treatment of Patients With Intra-abdominal Abscesses
Acronym: MEMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHH-MW-01
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Abscess, Intra-Abdominal
Keywords: abscess; intraabdominal abscess; Moxifloxacine; Moxifloxacin; Metronidazole; Tazobactam; Piperacilline; Piperacillin; Tazobac
MeSH Terms: conditions — Abdominal Abscess; Abscess | interventions — Moxifloxacin; Metronidazole; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): For adult patients with intra-abdominal abscesses matching the criteria to be included will and enrolled in the study arm 1: Moxifloxacin 400 mg, administered intravenously once daily in combination with Metronidazole 500 mg, administered two times daily intravenously, followed by an oral medication with Moxifloxacin 400 mg once daily and Metronidazole 500 mg twice daily.
  Interventions: Drug: Moxifloxacin/Metronidazole or Piperacillin/Tazobactam
- 2 (Active Comparator): For adult patients with intra-abdominal abscesses matching the criteria to be included will and enrolled in the study arm 2: Piperacillin / Tazobactam 4,5 g administered intravenously three times daily
  Interventions: Drug: Moxifloxacin/Metronidazole or Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Moxifloxacin/Metronidazole or Piperacillin/Tazobactam — Antibiotic therapy for patients with intra-abdominal abscesses; Intervention consists of antibiotic treatment of the patients with intraabdominal abscess with either the combination of Moxifloxacin and Metronidazole or Piperacillin/Tazobactam.1. Moxifloxacin 400 mg, administered intravenously once daily in combination with Metronidazole 500 mg, administered two times daily intravenously, followed by an oral medication with Moxifloxacin 400 mg once daily and Metronidazole 500 mg twice daily. 2. Piperacillin / Tazobactam 4,5 g administered intravenously three times daily.

SUMMARY:
The study is contemplating the antibiotic therapy of intraabdominal abscesses. These abscesses are a serious problem in surgical practice. Associated pathophysiologic effects as for example peritonitis may become life threatening or may lead to extended periods of morbidity with prolonged hospitalization.

The objective of the sudy is to evaluate whether the combination of Moxifloxacin and Metronidazole is equivalent to Piperacillin / Tazobactam with regard to clinical outcome and eradication of aerobe and anaerobe pathogens in patients with intra-abdominal abscesses.

DETAILED DESCRIPTION:
The study is an interventional prospective, comparative, open-label, randomised single-centre study. Adult patients with intra-abdominal abscesses matching the criteria to be included will be enrolled in the study and randomised into one of the Groups: 1. Moxifloxacin 400 mg, administered intravenously once daily in combination with Metronidazole 500 mg, administered two times daily intravenously, followed by an oral medication with Moxifloxacin 400 mg once daily and Metronidazole 500 mg twice daily. 2. Piperacillin / Tazobactam 4,5 g administered intravenously three times daily.

Primary study endpoints: Clinical success / failure rate at the Test-of-Cure visit.

Secondary study endpoints: -Bacteriological response at TOC, -Clinical + Bacteriological response at End-of-Treatment-visit, - Course of disease on the basis of clinical and laboratory parameters, -Time to discharge from hospitals, -Duration of hospitalization post-operatively, - safety and tolerability of the study medication, -cost effectiveness of treatment regimes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who attained full age (18 years) with intra-abdominal abscesses documented by:

A) Laparotomy revealing intra-abdominal abscess or macroscopic gastrointestinal perforation OR

B) Suspected intra-abdominal abscess and scheduled for operation with at least three of the following criteria:

* fever,
* leucocytosis,
* symptoms referable to the abdominal cavity (nausea, pain),
* tenderness with or without rebound / abdominal wall rigidity,
* radiological evidence for abscess or gastrointestinal perforation.

Exclusion Criteria:

* Patients with the following:

  * indwelling peritoneal catheter,
  * presumed spontaneous bacterial peritonits,
  * peripancreatic sepsis or infection secondary to pancreatitis,
  * peptic or traumatic perforation of gastrointestinal tract of < 24 h duration,
  * traumatic perforation of the small or large bowel of < 12h duration,
  * transmural necrosis of the intestine due to acute embolic, thrombotic or obstructive occlusions,
  * acute cholecystitis,
  * appendicitis without perforation or abscess,
  * required open abdomen techniques for management,
  * gynaecological infection,
  * known hypersensivity to any of the study drugs,
  * lifethreatening disease with life expectancy of less than 48 hours,
  * neutropenia with neutrophil count < 1000 cells/µl,
  * receiving chronic treatment with imunosuppressant therapy,
  * HIV-seropositives with CD4 count < 200 cells/µl,
  * end stage hepatic cirrhosis CHILD PUGH C,
  * central or peripheral neuropathy,
  * bradycardia,
  * symptomatic dysrhythmia in medical history,
  * syndromes of QTc prolongation or use of concomittant medicaments reported to increase QT interval,
  * disorder of the electrolyte balance,
  * previous history of tendinopathy with quinolones,
  * previously enrolled in the trial or use of any investigational drug within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-11-15 (Actual); Primary Completion 2011-08-15 (Actual); Study Completion 2011-08-15 (Actual)

PRIMARY OUTCOMES:
Clinical success / failure rate at the Test-of-Cure visit | 14 days
  clinical success

SECONDARY OUTCOMES:
Clinical + Bacteriological response at End-of-Treatment-visit | 14 days
  microbiology
Time to discharge from hospital | up to several months
  hospital stay
Course of disease on the basis of clinical and laboratory parameters | several days
  response to treatment
safety and tolerability of the study medication | 4 to 10 days
  recording of side effects od study medication such as cardiac arrythmias
cost effectiveness of treatment regimes | up to several months
  total costs of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Michael Winkler, Prof, Principal Investigator — Medical School Hannover, Department for abdominal and transplant surgery
Locations (1):
- Medical School Hannover, Hanover, Germany